CLINICAL TRIAL: NCT01539694
Title: A Study to Evaluate the Product Performance of a Low Add MultiFocal Soft Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: 744E
Record Dates: First submitted 2012-02-15; First posted 2012-02-27 (Estimated); Results first posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LD118033 contact lens (Experimental): Investigational LD118033 multifocal low add soft contact lenses, to be worn on a daily wear basis.
  Interventions: Device: LD118033 contact lens
- PureVision multifocal contact lens (Active Comparator): PureVision multifocal low add soft contact lens, to be worn on a daily wear basis.
  Interventions: Device: PureVision multifocal contact lens

INTERVENTIONS:
Device: LD118033 contact lens — Multifocal contact lens worn on a daily wear basis for 1 week
  Arms: LD118033 contact lens
Device: PureVision multifocal contact lens — PureVision multifocal contact lens worn on a daily wear basis for 1 week.
  Arms: PureVision multifocal contact lens

SUMMARY:
The objective of this study is to evaluate the product performance of an investigational multifocal low add soft contact lens.

ELIGIBILITY:
Inclusion Criteria:

* Have physiologically normal anterior segments.
* Be adapted wearers of soft contact lenses and wear a lens in each eye.
* Be presbyopic and require near add correction in each eye.
* Have no active ocular disease or allergic conjunctivitis.
* Must not be using any topical ocular medications.

Exclusion Criteria:

* Any Grade 2 or greater finding during the slit lamp examination.
* Any scar or neovascularization within the central 4mm of the cornea.
* Any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Allergic to any component in the study products.
* Any systemic disease affecting ocular health.
* Using any systemic or topical medications that will affect ocular physiology or lens performance.
* An active ocular disease, any corneal infiltrative response or are using any ocular medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Cairns, PhD, MCOptom, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 126 participants (252 eyes) were enrolled. One-half of the participants were randomized to receive the investigational contact lens during the first crossover period, and the other half were randomized to receive the PureVision contact lens during the first crossover period. The participants crossed over to the other group at 1 week.
Groups:
- LD118033 Contact Lens Then PureVision Multifocal Contact Lens: Investigational LD118033 multifocal low add soft contact lenses, to be worn on a daily wear basis.
  LD118033 contact lens: Multifocal contact lens worn on a daily wear basis for 1 week
  PureVision multifocal low add soft contact lens, to be worn on a daily wear basis.
  PureVision multifocal contact lens: PureVision multifocal contact lens worn on a daily wear basis for 1 week
- PureVision Multifocal Contact Lens Then LD118033 Contact Lens: PureVision multifocal low add soft contact lens, to be worn on a daily wear basis.
  PureVision multifocal contact lens: PureVision multifocal contact lens worn on a daily wear basis for 1 week.
  Investigational LD118033 multifocal low add soft contact lenses, to be worn on a daily wear basis.
  LD118033 contact lens: Multifocal contact lens worn on a daily wear basis for 1 week
Period: Overall Study
Arm/Group | LD118033 Contact Lens Then PureVision Multifocal Contact Lens | PureVision Multifocal Contact Lens Then LD118033 Contact Lens
Started | 63 | 63
Completed | 62 | 62
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Demography was collected for 124 eligible, dispensed participants. Participants received both treatment groups.
Groups:
- Overall: All participants/eyes received both treatment groups.
Arm/Group | Overall
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Visual acuity was assessed by distance high contrast logarithm of the minimum angle of resolution (logMAR).
Time Frame: At 1 week follow up
Population: There were 124 eligible, dispensed participants (248 eyes). Participants/eyes received both treatment groups.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | LD118033 Contact Lens | PureVision Multifocal Contact Lens
Number analyzed (Participants) | 124 | 124
Number analyzed (eyes) | 248 | 248
logMAR | 0.023 (0.078) | 0.005 (0.069)

2. Secondary Outcome: Symptoms/Complaints
Description: Symptoms/complaints were assessed on a scale from 0 to 100, with 0 denoting unfavorable symptoms/complaints.
Time Frame: At 1 week follow up
Population: There were 124 eligible, dispensed participants (248 eyes). Participants/eyes received both treatment groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | LD118033 Contact Lens | PureVision Multifocal Contact Lens
Number analyzed (Participants) | 124 | 124
Number analyzed (eyes) | 248 | 248
score on a scale
  Burning/stinging upon insertion | 91.3 (12.6) | 89.2 (16.9)
  Comfort upon insertion | 87.0 (16.6) | 83.9 (18.0)
  Comfort at end of day | 72.5 (24.4) | 68.1 (25.0)
  Overall comfort | 79.2 (21.2) | 74.6 (22.9)
  Dryness | 78.7 (22.4) | 75.2 (23.7)
  Itchiness | 89.1 (17.0) | 84.5 (21.1)
  Redness | 91.9 (12.3) | 87.0 (18.0)
  Distance Vision | 69.3 (30.4) | 76.5 (23.3)
  Vision at intermediate distance | 81.2 (20.3) | 80.7 (18.3)
  Vision at near distance | 76.3 (25.7) | 72.2 (26.2)
  Overall vision | 72.9 (25.8) | 73.7 (22.7)
  Ease of handling/insertion | 85.7 (18.8) | 85.4 (19.7)
  Ease of handling/removal | 88.5 (17.2) | 87.5 (17.5)
  Overall impression | 24.7 (24.0) | 74.6 (22.7)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Adverse events (AEs) were not coded. Therefore, source vocabulary is not applicable. A total of 126 participants (252 eyes) were assessed for AEs. Participants/eyes received both treatment groups in this cross-over study.
Arm/Group | LD118033 Contact Lens | PureVision Multifocal Contact Lens
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/126
Other Adverse Events (participants affected / at risk) | 0/126 | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.